CLINICAL TRIAL: NCT04942015
Title: Beijing University of Chinese Medicine
Brief Title: Honghuaruyi Wan for Endometriosis Dysmenorrhea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, mei han, Researcher, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HHRYW2021-05
Record Dates: First submitted 2021-05-27; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Endometriosis; Dysmenorrhea
MeSH Terms: conditions — Endometriosis; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honghuaruyi Wan (Experimental): Honghuaruyi Wan will be used in this arm. Patients should start taking medicine with warm water on the first day of menstruation. For patients with VAS score < 7 points, 1g / time, twice a day; for patients with VAS score ≥ 7 points and pain is hard to bear, 2g / time, twice a day. According to the above usage and dosage, take 3 menstrual cycles continuously, and observe 3 menstrual cycles after stopping the drug.
  Interventions: Drug: Honghuaruyi Wan
- Placebo (Placebo Comparator): Placebo of Honghuaruyi Wan will be used in this arm. Patients should start taking medicine with warm water on the first day of menstruation. For patients with VAS score < 7 points, 1g / time, twice a day; for patients with VAS score ≥ 7 points and pain is hard to bear, 2g / time, twice a day. According to the above usage and dosage, take 3 menstrual cycles continuously, and observe 3 menstrual cycles after stopping the drug.
  Interventions: Drug: Placebo of Honghuaruyi Wan

INTERVENTIONS:
Drug: Honghuaruyi Wan — Honghuaruyi Wan is the traditional Tibetan prescription, clinical research has proved that Honghuaruyi Wan can significantly reduce risk mouse dysmenorrhea caused by oxytocin, improve dysmenorrhea model of mice body torsion times and improve the estrogen and progestogen operator Netherlands rat pituitary estradiol and prolactin level, at the same time also can reduce the amount of TNF alpha, thus improving endometriosis dysmenorrhea.(Pill (15 pills/plate ×2 plates/box))
  Arms: Honghuaruyi Wan
Drug: Placebo of Honghuaruyi Wan — Honghuaruyi Wan simulation agent. Made of starch,dextrin and edible pigment from Tibet Qizheng Tibetan Medicine Co.,Ltd. ( Pill (15 pills/plate ×2 plates/box))
  Arms: Placebo

SUMMARY:
Endometriosis is a common gynecological disease. It is a gynecological disease caused by the growth and reproduction of the endometrium beyond the surface of the uterine tissue and organs, which causes recurrent abdominal pain, infertility and other main symptoms.

The recurrence of endometriosis and the side effects of medication have troubled clinicians and patients for a long time and the search for new drugs is going on all the time. Honghuaruyi Wan is the traditional Tibetan prescription, clinical research has proved that Honghuaruyi Wan can significantly reduce risk mouse dysmenorrhea caused by oxytocin, improve dysmenorrhea model of mice body torsion times and improve the estrogen and progestogen operator Netherlands rat pituitary estradiol and prolactin level, at the same time also can reduce the amount of TNF alpha, thus improving endometriosis dysmenorrhea.

In this study, the therapeutic effects of Honghuaruyi Wan provided by Tibet Qizheng Tibetan Medicine Co.,Ltd on secondary dysmenorrhea in patients with endometriosis was evaluated clinically. A multi-center, randomized, double-blind, placebo-controlled clinical trial was designed to provide evidence-based medical evidence for Honghuaruyi Wan in the treatment of endometriosis dysmenorrhea. In the design of this trial, the therapeutic effects and safety of Honghuaruyi Wan in the treatment of dysmenorrhea secondary to endometriosis were evaluated with Honghuaruyi Wan in the treatment group and placebo in the control group.

DETAILED DESCRIPTION:
Endometriosis (EM) is a common gynecological disease at present. It is a gynecological disease caused by the growth and reproduction of the endometrium on the surface of tissues and organs beyond the uterine covering surface, resulting in recurrent abdominal pain and infertility. The pathogenesis of endometriosis may be related to female endocrine dysfunction and abnormal levels of estrogen and progesterone in the body. Its clinical symptoms mainly include dysmenorrhea, chronic pelvic pain and sexual pain.

The recurrence of endometriosis and the side effects of medication have troubled clinicians and patients for a long time. The search for new drugs has been going on.

Honghuaruyi Wan is a traditional Tibetan prescription, which is made by addition and subtraction on the basis of the traditional and classic Tibetan medicine prescription "25 Wei Guijiu Wan". Its main ingredients are: Honghua,Xihonghua,Taoerqi,Kezi,Zangqiancao,Rougui,Baxiaga,Zangmuxiang,Yuansuiguo,Jiangxiang,Xiongdanfen,Zangzicao,Guangmingyan,Ximalayazimoli,Bangga,Hujiao,Huasherou,Aizijin,Yuganzi,Shajigao,Naosha,Zicaorong,Gouqizi,Chenxiang,Huoxiao. It has the effects of dispelling wind-evil and relieving pain, regulating menstrual blood and removing spots. It can be used for vaginitis, cervical erosion, irregular menstruation, dysmenorrhea and other common gynecological diseases. The main medicinal ingredients of Honghuaruyi Wan are Honghua ,Taoerqi and Zanghonghua, which have the effects of relieving pain, regulating menstruation and blood and dispersing knots. Some clinical studies have shown that the basic prescription of Honghuaruyi Wan have a significant effect on the improvement of dysmenorrhea, which can significantly reduce the incidence of dysmenorrhea caused by oxytocin in mice, and improve the number of body twisting in dysmenorrhea model mice. Other clinical studies have shown that Honghuaruyi Wan can improve estradiol and prolactin levels of pituitary gland in rats with estrogen and progesterone, as well as reduce TNF-α levels, thus improving endometriosis dysmenorrhea.

For women of childbearing age who do not have fertility requirements, pain is the most important clinical symptom that needs to be addressed, especially with progressive dysmenorrhea. Therefore, in this study, the therapeutic effects of Honghuaruyi Wan, provided by Tibet Qizheng Tibetan Medicine Co.,Ltd, on the secondary dysmenorrhea of patients with endometriosis was evaluated clinically. A multi-center, randomized, double-blind, placebo-controlled clinical trial was designed to provide evidence-based medical evidence for Honghuaruyi Wan in the treatment of endometriosis dysmenorrhea.

In the design of this trial, the therapeutic effects and safety of Honghuaruyi Wan in the treatment of dysmenorrhea secondary to endometriosis were evaluated with Honghuaruyi Wan in the treatment group and placebo in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for endometriosis and have dysmenorrhea VAS score ≥4 points;
2. Age 18 to 45;
3. Regular menstrual cycle (28±7 days);
4. Not pregnant at the time of seeing a doctor and no pregnancy plan during the medication, can insist on contraception;
5. No pelvic nodules or adnexal masses, or pelvic nodules or adnexal masses ≤4cm;
6. CA125 is normal or slightly elevated (below 200U/ml).
7. Patients who voluntarily signed the informed consent and had conditional follow-up.

Exclusion Criteria:

1. Patients who have known to have malignancies of reproductive organs or other malignancies;
2. Suffering from serious diseases or mental diseases such as cardiovascular, cerebrovascular, liver, kidney or hematopoietic system;
3. Uterine fibroids (≥3cm) and adenomyosis (uterine over 6 weeks of gestation, the reference value of uterine tridiameter at 6 weeks is 12cm, 7.5cm, 4.5cm);
4. Those who received hormone drug therapy within 3 months before enrollment;
5. lactating patients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-06-21 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale/Score (VAS) | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  Draw a horizontal line of 10 cm on the paper. One end of the horizontal line is 0, indicating no pain.The other end is 10, which means severe pain; The part between the two ends represents different levels of pain. A higher score means a worse outcome.
Endometriosis Health Profle-5（EHP-5） | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  The core questionnaire contains 5 questions，every question has 5 answers：Never=0，Very few=1，Sometimes=2，Often=3，Always=4. The minimum and maximum values are between 0 to 20 and a higher value means a worse outcome.
The 5-level EQ-5D version（EQ-5D-5L） | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  There are 6 questions in the scale，the first 5 questions has 5 answers：No=0， A little bit=1， Moderate=2， Serious=3 Very serious=4. The minimum and maximum values are between 0 to 20 and a higher value means a worse outcome. The 6th question is about the status of the day visited. The minimum and maximum scores are between 0 to 100 and a higher value means a better outcome.

SECONDARY OUTCOMES:
Visual Analogue Scale/Score (VAS) of the maximum non-menstrual pelvic pain | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  Draw a horizontal line of 10 cm on the paper. One end of the horizontal line is 0, indicating no pain.The other end is 10, which means severe pain; The part between the two ends represents different levels of pain. A higher score means a worse outcome.
The number of ibuprofen sustained-release capsules (or other NSAIDs) used | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  The number of ibuprofen sustained-release capsules (or other NSAIDs) used
Number of days off for staff/students due to dysmenorrhea | Baseline through 6th consecutive menstrual cycle. (One cycle = 28±7days)
  Number of days off for staff/students due to dysmenorrhea
The maximum diameter of the uterus | Baseline, After treatment (3rd menstrual cycle). (One cycle = 28±7days)
  The diameter of the uterus will be measured by B ultrasonic
The maximum diameter of the cysts | Baseline, After treatment (3rd menstrual cycle). (One cycle = 28±7days)
  The diameter of the cysts will be measured by B ultrasonic

CONTACTS AND LOCATIONS:
Overall Officials: Mei Han, Study Chair — Centre for Evidence-based Chinese Medicine, Beijing University of Chinese Medicne

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are limited upon to contract with the company and might be made available upon agreement from the company.

REFERENCES:
- [Derived] Han M, Liang XF, Gao J, Wang Y, Cao LX, Wang BJ, Wang Y, Zhuoma Z, Liu JP, Du HL. Honghua Ruyi Pill, a compound herbal medicine, improves endometriosis-related dysmenorrhea: A multicenter randomized, double-blind, placebo-controlled trial. J Integr Med. 2025 Dec 29:S2095-4964(25)00203-1. doi: 10.1016/j.joim.2025.12.011. Online ahead of print. PMID 41529972